CLINICAL TRIAL: NCT04794920
Title: Post-Covid-19 Emotional Aspects of Hospital Staff
Acronym: EMOCOV
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: EMOCOV
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Covid19
Keywords: Emotional aspects; caregivers
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ongoing SARS-CoV2 or Covid-19 pandemic is causing a major global health crisis. In France, it prompted an urgent reorganization of the healthcare supply, mobilizing caregivers and hospital staff in a climate of uncertainty. Health services have been put to the test, some staff being on the front line, others having faced the reorganization of the health system necessitated by such a pandemic.

Frontline caregivers have been compared to "fighters on the front lines." They encountered many difficulties, such as direct exposure to patients with a high viral load, exposure to the risk of contamination, physical exhaustion, reorganization of workspaces, adaptation to rigid work organizations, the management of the shortage of materials, the unusually high number of deaths among patients, colleagues or relatives, ethical questions relating to decision-making in a strained healthcare system.

The psychological impact on these hospital staff is an indirect issue of such a pandemic in terms of mental health.

The investigators have little data in the literature on the incidence of psychiatric episodes in the post-epidemic period. Work on the impact of two major pandemics of influenza A H1N1 (2009) and SARS-CoV-1 (2003) on the mental health of caregivers and other staff working in hospitals reports increased rates of mental disorders after discharge from anxiety-type crisis, depression and post-traumatic stress. This over-representation of mental disorders was still found several years after the epidemic.

Similar results are emerging in recent studies involving hospital staff who were used in the Covid-19 crisis. These highlight a certain number of risk factors for the occurrence of these disorders (young age, nursing profession, underlying psychiatric pathology, exercise carried out in the first line of Covid).

DETAILED DESCRIPTION:
At the Paris Saint-Joseph Hospital Group (GHPSJ), a multidisciplinary working group was early involved in psychological support for staff.

This group proposed the establishment of on-call duty entrusted to a psychological support unit, made up of a doctor, a nurse and a psychologist who volunteered to carry out patrols in the various departments of the hospital. These visits, sometimes organized at the request of the management of the services and sometimes improvised, aimed to identify the difficulties encountered in the field, and to discuss with the teams.

Concomitantly and complementary, the staff bubble opened at the Paris Saint-Joseph Hospital on March 27, to offer a decompression space to all staff (caregivers or not) with proposals for hypnosis, physiotherapy, sophrology sessions. , psychotherapy, but also informal discussions or a break in a relaxing armchair.

As a continuation of this approach, the multidisciplinary working group plans to search in July 2020 for symptoms present in certain mental illnesses (anxiety, depression, post-traumatic stress syndrome) in all the staff of the Paris Saint-Joseph Hospital Group. , now that the crisis seems to be receding. This will make it possible to adapt the support offer for staff in the coming months. This inventory will be made on the basis of validated questionnaires: the Posttraumatic stress disorder CheckList-5 (PCL) questionnaire for post-traumatic stress and the Hospital Anxiety and Depression scale (HAD) score for mental disorders (anxiety, depression) . A 3rd questionnaire will collect additional data and provide feedback on the frequentation of the bubble

ELIGIBILITY:
Inclusion Criteria:

- Any staff (caregivers and non-carers) who worked during the Covid 19 crisis (from March 15 to May 15) at the GHPSJ, on site or by teleworking, all or part of the period.

Exclusion Criteria:

- Opposition to participate in research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any staff (caregivers and non-carers) who worked during the Covid 19 crisis (from March 15 to May 15) at the GHPSJ, on site or by teleworking, all or part of the period
Sampling Method: Non-Probability Sample
Enrollment: 780 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2020-10-03 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Frequency of symptoms related to post-traumatic stress in all staff who worked at the GHPSJ during the crisis (from March 15 to May 15, 2020). | Day 1
  Rate of staff with a score> 44 on the PCL questionnaire
Frequency of symptoms related to post-traumatic stress in all staff who worked at the GHPSJ during the crisis (from March 15 to May 15, 2020). | Day 1
  Rate of staff with a score ≥11 on items A and D for the HAD score

SECONDARY OUTCOMES:
Look for demographic and professional characteristics that may favor the onset of these symptoms | Day 1
  Univariate and multivariate analyzes to identify the risk factors for the occurrence of these symptoms (anxiety, depression and post-traumatic stress)
Evaluate the impact of frequentation of the staff bubble on the occurrence of anxiety / depressive disorders | Day 1
  Difference between the average HAD scores between the group "frequentation of the staff bubble" and the group "non-attendance of the staff bubble". The distinction between the 2 groups is made on the basis of their answer to the dedicated question asked in the questionnaire.
Evaluate the impact of frequentation of the staff bubble on the occurrence of post-traumatic stress | Day 1
  Difference between the mean PCL scores between the 2 above-mentioned groups
Evaluate the impact of the psychological support unit on the occurrence of anxiety / depressive disorders | Day 1
  Difference between the average HAD scores between the "contact with the psychological support unit" group and the "no contact with the psychological support unit" group. The distinction between the 2 groups is made on the basis of their response to the question asked in the questionnaire.
Evaluate the impact of the psychological support unit on the occurrence of post traumatic stress | Day 1
  Difference between the mean PCL scores between the 2 above-mentioned groups
Evaluate the benefit felt by staff from frequenting the staff bubble | Day 1
  In the group "frequentation of the staff bubble": percentage of response "Very beneficial" or "Quite beneficial"
Evaluate the benefit felt by the staff of the meeting with the psychological support unit | Day 1
  In the group "meeting with the psychological support unit": percentage of response "Very beneficial" or "Quite beneficial"

CONTACTS AND LOCATIONS:
Overall Officials: Marguerite D'USSEL, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, Île-de-France Region, France

REFERENCES:
- [Result] d'Ussel M, Fels A, Durand X, Lemogne C, Chatellier G, Castreau N, Adam F. Factors associated with psychological symptoms in hospital workers of a French hospital during the COVID-19 pandemic: Lessons from the first wave. PLoS One. 2022 Apr 28;17(4):e0267032. doi: 10.1371/journal.pone.0267032. eCollection 2022. PMID 35482772